CLINICAL TRIAL: NCT00295438
Title: Robot-based Tele-echography II - A Comparative Study Using Two Echographic Modalities for Diagnosis of Thoracoabdominal Injuries at the Trauma Center of the Grenoble University Hospital.
Brief Title: Robot-based Tele-echography II - A Comparative Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No diagnosis of visceral lesion was placed on 18 included patients. The study is thus stopped prematurely for ethical reasons.
Sponsor: University Hospital, Grenoble (Other)
Collaborators: France Telecom R&D (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 05 52
Record Dates: First submitted 2006-02-21; First posted 2006-02-23 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Abdominal Injuries; Thoracic Injuries; High Energy Trauma
Keywords: robot-based tele-echography; tele-medicine
MeSH Terms: conditions — Abdominal Injuries; Thoracic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot-Based Tele-Echography (TER) (Experimental): ultrasound performed according to the method Tele-Echography
  Interventions: Device: Robot-Based Tele-Echography (TER); Device: ultrasound method FAST
- ultrasound method FAST (Active Comparator): ultrasound performed according to the method FAST (Focused Assessment Sonography for Trauma)
  Interventions: Device: Robot-Based Tele-Echography (TER); Device: ultrasound method FAST

INTERVENTIONS:
Device: Robot-Based Tele-Echography (TER) — Robot-Based Tele-Echography, ultrasound performed by the radiologist
Device: ultrasound method FAST — FAST,ultrasound performed by the emergency doctor

SUMMARY:
The aim of this clinical trial is to evaluate the concordance of diagnosis of injuries in thoracoabdominal trauma using two different echographic methods. The first method is a robot-based tele-echography performed by radiologists in a remote location. The second is bedside echography performed by emergency physicians according to the FAST (Focussed Assessment by Sonography of Trauma) examination.

DETAILED DESCRIPTION:
1. Principal objective: to evaluate the concordance of diagnosis of injuries in thoracoabdominal trauma using two different echographic methods (robot-based tele-echography performed by radiologists in a remote location vs bedside echography performed by emergency physicians according to the FAST examination).
2. Objective 2: after the realization of a gold standard method, if there is a concordance between the two different echographic methods, sensitivity and specificity are estimated. If not, the evaluation of sensitivity and specificity of each method with analysis of their discordance is performed.
3. Objective 3: qualitative evaluation of each echographic method by the patient and the physicians.
4. Material and methods: This therapeutic, mono-centre, prospective, randomized, cross-over, open, controlled trial is being conducted in 70 patients. All the patients will have the two different echographic methods in a sequential but randomized way. The robot-based tele-echography is performed by a radiologist in the North University Hospital of Grenoble. The bedside echography is performed by the emergency physicians in the trauma center in the South University Hospital of Grenoble.

ELIGIBILITY:
Inclusion Criteria:

* Person registered with the French Social Security or benefiting from an equivalent health insurance system
* Person sent to hospital for thoracoabdominal high energy trauma

Exclusion Criteria:

* Ward of court or under guardianship
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Person participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-02; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The diagnosis concordance between the radiologists using the robot-based tele-echography and the emergency physicians (FAST bedside examination) is evaluated thanks to the Cohen kappa interrater agreement coefficient. | 6 month

SECONDARY OUTCOMES:
sensitivity, specificity, PPV, NPV are estimated with a 95% confidence interval | 6 month
qualitative scores (including comfort and experience of the patient, quality of the echographic method evaluated by the physicians). | 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Banihachemi, MD, Principal Investigator — Urgences Traumatologiques de l'hôpital SUD - Centre Hospitalier et Universitaire - Grenoble - B.P. 185 38042 GRENOBLE Cedex 09 - France
Locations (1):
- University Hospital, Grenoble, France

REFERENCES:
- [Background] Vilchis A, Masuda K, Troccaz J, Cinquin P. Robot-based tele-echography: the TER system. Stud Health Technol Inform. 2003;95:212-7. PMID 14663989